CLINICAL TRIAL: NCT05274347
Title: A Virtual Post-Discharge Intervention to Prevent Hospital Re-Admissions in Patients With CKD
Brief Title: A Virtual Post-Discharge Intervention For Patients With CKD
Acronym: VIDIO-CKD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14620
Record Dates: First submitted 2022-02-14; First posted 2022-03-10 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-faceted virtual, remote intervention (Experimental): The intervention will use the Aetonix - aTouchAwayTM software platform (AETONIX Systems Inc). Each study participant will receive a tablet with Aetonix software. Interventions Components:
  1. Cognitive behavioral therapy (CBT): After discharge, patients will receive weekly group CBT sessions delivered virtually by a psychologist. Throughout the series of CBT sessions, patients will learn strategies for problem-solving, assertive communication, relaxation, behavioural activation, time-based pacing, challenging unhelpful thinking, building motivation, and goal setting.
  2. Remote monitoring of vital signs and symptoms: Messages will be sent to patients asking them to measure their vitals, to report symptoms, and answer questions about medications. Concerning responses will be flagged for review by the patient's healthcare team.
  Interventions: Other: Muti-faceted virtual, remote intervention

INTERVENTIONS:
Other: Muti-faceted virtual, remote intervention — Patients will be provided with tablets with internet connectivity and Aetonix software, along with a blood pressure cuff, weigh scale and pulse oximeter with blue tooth capability. These will be used to deliver virtual CBT sessions as well as remote monitoring of vital signs, symptoms and enhanced communication. The intervention duration will be 10 weeks.

SUMMARY:
This pilot, interventional study is testing a combination of remote, virtual interventions, delivered to patients at home to patients with chronic kidney disease (CKD), with the goal of reducing admissions to hospital.

DETAILED DESCRIPTION:
Chronic kidney disease and kidney failure increase the risk of hospitalizations. Many hospital admissions are potentially avoidable. This pilot, interventional study is testing a combination of remote, virtual interventions, delivered to patients at home, with the goal of reducing admissions to hospital. The hypothesis for this pilot work is that the proposed interventions will be adopted by patients and will improve mental health, physical function, quality of life, and disease self-management, which are all key potential mediators of hospital readmission risk in patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults with CKD (defined as an estimated glomerular filtration rate <30mL/min/1.73m2, including hemodialysis)
* Able to provide informed consent.
* Ongoing follow-up by the St Joseph's Hospital Hamilton Kidney Care Clinic or Dialysis Program and with a recent hospital admission.

Exclusion Criteria:

* Unable to speak or understand English.
* Significant cognitive impairment (as per the treating inpatient care team)
* Serious mental illness (schizophrenia, severe untreated bipolar disorder, psychosis, active suicidal ideation)
* Significant vision or hearing impairment that prevents use of the technology or participation in any of the intervention components.
* Being discharged to long-term care, rehab or complex care.
* Peritoneal dialysis
* Home hemodialysis
* Functioning kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Patient uptake of the intervention | 10 weeks
  Patient use of the Aetonix platform and virtual intervention components. Uptake of the virtual CBT intervention will be determined by the number of attended sessions.
Patient acceptance of the intervention | 10 weeks
  Acceptability of the technology will be determined by the proportion of patients who provide a mean Telehealth Usability Questionnaire (TUQ) score >5/7. The mean TUQ score ranges from 1 to 7, with a higher score indicating greater acceptance of the intervention.

SECONDARY OUTCOMES:
Patients' reasons for not participating in virtual sessions. | 10 weeks
  This will be collected for further detail on the uptake of the intervention.
Patient satisfaction with the intervention | Measured at 10 weeks (study end)
  Satisfaction with both the technology and virtual physiotherapy and CBT sessions. This outcome will be determined using a locally developed patient experience survey instrument that includes 13 questions asking patients to rate various elements of the intervention with the response options "strongly disagree", "disagree", "neutral", "agree", "strongly agree". The Satisfaction with Therapy and Therapist Scale- Revised (STTS-R) will be used to measure satisfaction with the CBT intervention.
Uptake of systolic and diastolic blood pressure monitoring | 10 weeks
  Mean number of missing blood pressure values per patient.
Changes in management as a result of remote monitoring | 10 weeks
  Mean number of alert values per patient from the monitoring pathway, mean number of alerts that resulted in a change in management per patient, mean number of medication errors detected per patient
Change in depression | 10 weeks
  Change in Patient Health Questionnaire-9 (PHQ-9) score (measured every 2 weeks). The PHQ-9 score ranges from 0 to 27. A higher score indicates a higher degree of depressive symptoms.
Change in anxiety | 10 weeks
  Change in Generalized Anxiety Disorder-7 (GAD-7) score (measured every 2 weeks). The GAD-7 score ranges from 0 to 21, with a higher score indicating a higher degree of anxiety.
Change in disease self-efficacy | 10 weeks
  Change in Self Efficacy for Managing Chronic Disease (SEMCD) score (measured every 2 weeks). The SEMCD score is the mean score from 6 items, with a means score range from 1 to 10. A higher score indicates higher self-efficacy
Change in overall self-reported health | 10 weeks
  Measured every 2 weeks using the single question Global QOL score. Participants will be asked to rate their overall health as "excellent, good, fair, or poor".
Change in self-reported quality of life | 10 weeks
  measured week 1, week 5 and week 10 using the Short Form-36 (SF-36) questionnaire. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability
Questionnaire completion | 10 weeks
  Mean number of incomplete questionnaires per patient
All-cause hospitalizations | 10 weeks
  Hospitalizations will be determined by patient report directly into their Aetonix tablet (weekly question) or clinical staff following up on alerts for missed CBT/physio sessions or >3 consecutive missed daily symptom/vitals questionnaires.
Emergency room visits | 10 weeks
  Emergency room visits will be determined by patient report directly into their Aetonix tablet (weekly question) or clinical staff following up on alerts for missed CBT/physio sessions or >3 consecutive missed daily symptom/vitals questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Amber O Molnar, MD, MSc, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No